CLINICAL TRIAL: NCT05131100
Title: Korean Post-marketing Surveillance for Somavert
Brief Title: Korean Regulatory Post Marketing Surveillance for Somavert
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6291047; NCT05131100 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2021-11-10; First posted 2021-11-23 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Acromegaly
Keywords: acromegaly, Somavert, Post-Marketing Surveillance
MeSH Terms: conditions — Acromegaly | interventions — pegvisomant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants receiving Somavert
  Interventions: Drug: Somavert

INTERVENTIONS:
Drug: Somavert — As provided in real world practice

SUMMARY:
Non-interventional observational study, to identify safety and effectiveness of Somavert during the post-marketing period based on the Korean RMP as required by the regulations of Ministry of Food and Drug Safety (MFDS)

ELIGIBILITY:
Inclusion Criteria:

All patients who have been prescribed as per local label and investigators' judgement under the setting of routine practice in Korea who are eligible.

Exclusion Criteria:

Patients who are contraindicated for Somavert

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult acromegaly patients who have had an inadequate response to surgery and/or radiation therapy and in whom appropriate medical treatment with somatostatin analogues did not normalize IGF-1 concentrations or was not tolerated
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience adverse events | Baseline through 28 days after last dose (approximately 52 weeks)

SECONDARY OUTCOMES:
Number of participants who experience Clinical Improvement as assessed by investigator | Baseline through approximately 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A6291047